CLINICAL TRIAL: NCT04590638
Title: Comparison Between Effect of Adrenaline and Without Adrenaline in Tumescent Solutions on Bleeding Control of Skin Graft Donor Site.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Principal Investigator, Mahak Ali, MahakA, Dow University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Mmehak
Record Dates: First submitted 2020-10-11; First posted 2020-10-19 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Bleeding Time
MeSH Terms: interventions — Epinephrine

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tumescent with adrenaline (Active Comparator): skin graft donor site of patients recurited in this group will be injected subcutaneously with tumescent solution containing adrenaline.
  Interventions: Other: tumescent with adrenaline
- Tumescent without adrenaline (Active Comparator): skin graft donor site of patients recurited in this group will be injected subcutaneously with tumescent solution not containing adrenaline.
  Interventions: Other: tumescent without adrenaline

INTERVENTIONS:
Other: tumescent with adrenaline — skin graft donor site of patients enrolled in this group will be injected subcutaneously with tumescent solution containing adrenaline to see the bleeding control of donor site.
  Arms: Tumescent with adrenaline
Other: tumescent without adrenaline — skin graft donor site of patients enrolled in this group will be injected subcutaneously with tumescent solution not containing adrenaline to see the bleeding control of donor site.
  Arms: Tumescent without adrenaline

SUMMARY:
The purpose of this study is to appraise if various concentration of adrenaline containing tumescent has any significant role in bleeding at skin graft donor site bleeding through photographic assessment.

DETAILED DESCRIPTION:
Tumescent solutions will be prepared by adding 30cc of Ringer's lactate and 10cc of lignocaine 2%, with 1cc of adrenaline of 1:200,000 (which will be prepared by adding 1cc of adrenaline of 1:1000 conc. with 200ml of normal saline marked as solution "A" and without adrenaline marked as solution "B" to form the two different tumescent solutions. Both solutions with be topically applied in soaked gauzes for around 10 minutes. Solution A will be applied over the anterior side of thigh while solution B will be applied over lateral side of thigh.

Tumescent solutions will be prepared around 10 minutes before applying. After 10 min Split-thickness skin graft donor sites will be harvested with a Dermatome adjusted on with a randomized setting to harvest a fixed depth of wound depth. After harvesting skin graft the donor site wound will be photographed.

The apparent severity of bleeding will be scored on an ordinal scale from 0 to 5 (0=no bleeding/staining, 1=minimal bleeding/staining, 2=mild bleeding/staining, 3=moderate bleeding/staining, 4=moderately severe bleeding/staining, 5=severe bleeding/staining by two independent surgeons. At last photographs will be compared with pre-infiltration records in each side. Skin graft donor and recipient site will be inspected on the 5th post-operative day

ELIGIBILITY:
Inclusion Criteria:

* age above 18 years

  * both genders
  * non hypertensive patients
  * Hemoglobin levels more than 10 g/dl
  * Platelet count above 150 x 10E9/L
  * Wounds for more than 6 weeks

Exclusion Criteria:

* • Hypertensive patients,

  * Bleeding tendencies (Disorder),
  * Immune-compromised,
  * Familial history of bleeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2020-10-17 (Actual); Primary Completion 2021-03-17 (Actual); Study Completion 2021-03-17 (Actual)

PRIMARY OUTCOMES:
ordinal scale | 30minutes
  The apparent severity of bleeding will be scored on an ordinal scale from 0 to 5 (0=no bleeding/staining, 1=minimal bleeding/staining, 2=mild bleeding/staining, 3=moderate bleeding/staining, 4=moderately severe bleeding/staining, 5=severe bleeding/staining by two independent surgeons.

CONTACTS AND LOCATIONS:
Locations (1):
- Mahak, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No